CLINICAL TRIAL: NCT03437876
Title: A Randomised Study on Intestinal Microbiota Transplantation for Hepatitis B Virus Induced Cirrhosis
Brief Title: Study on Effect of Intestinal Microbiota Transplantation in Hepatitis B Virus Induced Cirrhosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhongshan Hospital Xiamen University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2017002
Record Dates: First submitted 2017-10-25; First posted 2018-02-19 (Actual); Last update posted 2018-02-19 (Actual); Status verified 2017-10

CONDITIONS: Cirrhosis, Liver
Keywords: HBV induced cirrhosis; intestinal microbiota transplantation; microbiota
MeSH Terms: conditions — Liver Cirrhosis | interventions — Fecal Microbiota Transplantation

STUDY DESIGN:
Intervention Model Description: a open-label, self-control study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- patients with HBV induced cirrhosis (Experimental): patients with HBV induced cirrhosis will be recruited for study, which involved a 4 times intestinal microbiota transplant and the time interval is generally 2 weeks.
  Interventions: Other: intestinal microbiota transplant

INTERVENTIONS:
Other: intestinal microbiota transplant — All participants take 4 times IMT by gastroduodenoscopy with 2-week intervals

SUMMARY:
Chronic hepatitis B (CHB) is a common infectious disease affecting up to 2 billion people worldwide. Around 650 thousand people died of liver failure, cirrhosis and primary liver cancer caused by chronic hepatitis B every year. 3%-5% compensatory liver cirrhosis develop to decompensated cirrhosis and suffer from series symptoms such as fatigue, edema, portal hypertension, splenomegaly, hemorrhage, hepatic encephalopathy, hepatorenal syndrome and so on. Chronic hepatitis B is closely related to the imbalance of intestinal microbiota, and the intestinal microbiota of patients is significantly different from healthy people. The response of patients to hepatitis B virus can be influenced by reconstructing intestinal flora, while Intestinal microbiota transplantation(IMT) is a significant method to achieve it. In a previous study using IMT to treat HBeAg positive chronic hepatitis B patients combined with antiviral therapy, 80% of them has reached HBeAg clearance. The investigators propose a randomized trial of IMT in patients with HBV induced cirrhosis. Patients will be randomized to either control group or IMT group over a 12 months period.

DETAILED DESCRIPTION:
A group of 60 patients with HBV induced cirrhosis will be recruited for study, which involved a 4 times IMT with gastroduodenoscopy and the time interval is generally 2 weeks. Participants can keep taking their present treatment. All participants will be assessed at baseline, after 3 months, 6 months, 12 months from baseline in order to evaluate the possible changes in:

(1)Imaging changes: Color Doppler ultrasound of portal vein, CT/MRI, Fibroscan score of liver fibrosis and steatosis, Grading of varicosity under gastroscopy(GI); (2)Basic information and symptoms; (3)Biochemical indexes: Liver function, four items of liver fiber, lipid metabolism, blood routine, coagulation function, blood ammonia, inflammation, oxidative stress, urine routine; sugar metabolism indicators (blood glucose, glycosylated hemoglobin, insulin level and insulin resistance level).

(4) Changes of gut microbiota: The changes of gut microbiota will be assessed by High-throughput sequencing (16S rRNA) on baseline, 3 months, 6 months and 12 months after treatment samples to assess changes associated with IMT.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent/assent as appropriate, able to keep treatment
* 18 to 50 years of age
* Chronic hepatitis B, definitely diagnosed as hepatic fibrosis/cirrhosis through Fibroscan/Biopsy of liver biopsy

Exclusion Criteria:

* Drug treatment(immunosuppressive drugs, biological agents, high dose vitamins or other immunosuppressive drugs
* Other immune related diseases
* Gastrointestinal organic lesions such as gastroesophageal reflux disease, inflammatory bowel disease, intestinal tumor
* Medical or social condition which in the opinion of the principal investigator would interfere with or prevent regular follow up
* Participating in other clinical trials

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2016-10-31 (Actual); Primary Completion 2020-11 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
change of liver Fibroscan score | 3 months, 6 months, 12months
  Fibroscan score of liver fibrosis and steatosis

SECONDARY OUTCOMES:
Symptoms | 3 months, 6 months, 12months
  The onset and duration of gastrointestinal symptoms will be assessed by "Evaluation Score Table of Gastrointestinal Symptoms".
Changes of gut microbiota | 3 months, 6 months, 12months
  The changes of gut microbiota will be assessed by High-throughput sequencing (16S rRNA) in fecal samples from recruited patients.
Color Doppler ultrasound of portal vein | 3 months, 6 months, 12months
  Doppler ultrasonography is medical ultrasonography that employs the Doppler effect to generate imaging of the movement of tissues and body fluids (usually blood), and their relative velocity to the probe. By calculating the frequency shift of a particular sample volume, for example flow in an artery or a jet of blood flow over a heart valve, its speed and direction can be determined and visualized. Color Doppler is the presentation of the velocity by color scale. Color Doppler images are generally combined with grayscale (B-mode) images to display duplex ultrasonography images, allowing for simultaneous visualization of the anatomy of the area. This is particularly useful in cardiovascular studies (sonography of the vascular system and heart) and essential in many areas such as determining reverse blood flow in the liver vasculature in portal hypertension.
CT | 3 months, 6 months, 12months
  A CT scan, also known as computed tomography scan, makes use of computer-processed combinations of many X-ray measurements taken from different angles to produce cross-sectional (tomographic) images (virtual "slices") of specific areas of a scanned object, allowing the user to see inside the object without cutting. Other terms include computed axial tomography (CAT scan) and computer aided tomography.
MRI | 3 months, 6 months, 12months
  Hepatobiliary MR is used to detect and characterize lesions of the liver, pancreas, and bile ducts. Focal or diffuse disorders of the liver may be evaluated using diffusion-weighted, opposed-phase imaging, and dynamic contrast enhancement sequences. Extracellular contrast agents are used widely in liver MRI and newer hepatobiliary contrast agents also provide the opportunity to perform functional biliary imaging.

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongshan Hospital Affiliated to Xiamen University, Xiamen, Fujian, China

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (2):
  • Informed Consent Form (2017-06-28): https://cdn.clinicaltrials.gov/large-docs/76/NCT03437876/ICF_000.pdf
  • Study Protocol (2017-06-28): https://cdn.clinicaltrials.gov/large-docs/76/NCT03437876/Prot_001.pdf